CLINICAL TRIAL: NCT05021549
Title: Effectiveness of Apneic Oxygenation for Morbid Obese Parturient Performing Elective Caesarean Section Under General Anesthesia
Brief Title: Apneic Oxygenation for Morbid Obese Parturient in cs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Wael Elswefi, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: morbid obese parturient
Record Dates: First submitted 2021-08-20; First posted 2021-08-25 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: 1. Morbid obesity parturient defined as a body mass index (BMI) above 40 kg/m2.
  2. ASA physical status I-II
  3. Age above 18 years.
  4. Scheduled for elective caesarean section under general anesthesia.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nasal prong. (Active Comparator): the apneic preoxygenation group (30 patients), will receive 10 L/ min of O2 via nasal prong.
  Interventions: Device: nasal prong
- conventional (No Intervention): the conventional preoxygenation group (30 patients)

INTERVENTIONS:
Device: nasal prong — apneic preoxygenation group (30 patients), will receive 10 L/ min of O2 via nasal prong during preintubation apnia
  Arms: nasal prong.

SUMMARY:
The aim of this study is to compare the effect of apneic preoxygenation to conventional preoxygenation on the oxygen desaturation in morbid obese parturient performing elective caesarean section under general anesthesia.

DETAILED DESCRIPTION:
Anesthetic management of the obese parturient is challenging. Both pregnancy and obesity are risk factors for a difficult airway and anesthesia-related maternal mortality. There is increased risk of difficult intubation associated with an increased difficultly in mask ventilation and increased risk of accelerated desaturation during apnea.

The use of apneic oxygenation for the optimization of peri-intubation conditions is a promising means of preventing hypoxemia.

Despite the recommendation of the use of nasal prongs to insufflate oxygen at flows of 5 L/min to 15 L/min during the apneic period randomized controlled trial is still not available in the morbidly obese parturient.

ELIGIBILITY:
Inclusion Criteria:

1. Morbid obesity parturient defined as a body mass index (BMI) above 40 kg/m2.
2. ASA physical status I-II
3. Age above 18 years.
4. Scheduled for elective caesarean section under general anesthesia.

Exclusion Criteria:

1. Parturient of ASA physical status III or above.
2. Suspected or known difficult airway (Mallampati class > 2, reduced neck movement, reduced mouth opening, or Cormack-Lehane grade 4 recorded during a previous intubation procedure).
3. Any contraindication for nasal prong use, for example, tumours, fractures or trauma.
4. SpO2 ≤ 97% prior to preoxygenation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
the lowest oxygen saturation recorded | during intubation procedure
  percentage

SECONDARY OUTCOMES:
rates of desaturation below SpO2 90% | during intubation procedure
  percentage
rates of critical desaturation below SpO2 80% | during intubation procedure
  percentage

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ain Shams university, Cairo
  - Faculty of medicine, Cairo

IPD SHARING:
Plan to Share IPD: Yes
all IPD to be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after finishing the study
Access Criteria: clinicaltrial web site